CLINICAL TRIAL: NCT04578431
Title: Artificial Sweeteners in Breast Milk: A Clinical Investigation With a Kinetic Perspective
Brief Title: Artificial Sweeteners in Breast Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AS0063221
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2020-10

CONDITIONS: Breastfeeding; Diabetes Mellitus; Overweight
Keywords: Artificial sweeteners; Non-nutritive sweeteners
MeSH Terms: conditions — Breast Feeding; Diabetes Mellitus; Overweight | interventions — Sweetening Agents; acetosulfame; trichlorosucrose; Cyclamates

STUDY DESIGN:
Intervention Model Description: 60 women will be divided into three groups (n=20 each) based on pre-pregnancy BMI and metabolic status.
  The groups are
  1. Normal weight (BMI < 25),
  2. Over weight (BMI > 27),
  3. Diabetic
Masking Description: All participants are given the same intervention and are aware of this
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention groups (Experimental): The participants will be given a beverage containing four artificial sweeteners (intervention) at baseline
  Interventions: Dietary Supplement: Artificial sweeteners (acesulfame-potassium, sucralose, saccharine, cyclamate)

INTERVENTIONS:
Dietary Supplement: Artificial sweeteners (acesulfame-potassium, sucralose, saccharine, cyclamate) — The intervention is found in light products ingested by millions of people on a daily basis worldwide

SUMMARY:
This study will investigate how some artificial sweeteners (AS) cross from blood to breastmilk in breastfeeding women after oral intake. Moreover, it will be investigated whether the kinetics of AS differ based on the women's body composition (BMI) and metabolic status (diabetes). This will be investigated through a clinical trial in which 60 women divided into three groups (normal weight, overweight and diabetic) will drink a beverage containing four AS. over a period of six hours the women will donate blood and breast milk samples in order to investigate the presence of AS.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Able to give consent
* Able to produce enough amounts of breastmilk
* Danish/English speakers
* Pre-pregnancy BMI below 25 (20 subjects)
* Pre-pregnancy BMI above 27 (20 subjects)
* Diabetes type 1 or 2 (20 subjects)

Exclusion Criteria:

* Under the age of 18 years old
* Unable to give consent
* Unable to produce enough amounts of breastmilk
* Non-Danish/English speakers
* If they have consumed artificial sweeteners 24 hours prior to trial

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Breastmilk from mother | Baseline, after 30 mins and afterwards once and hour for six hours
  Concentration of artificial sweeteners in mother's breast milk
Blood from mother | Baseline, after 30 mins and afterwards once and hour for six hours
  Concentration of artificial sweeteners in mother's blood

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No